CLINICAL TRIAL: NCT02515682
Title: Effect of Natural S-equol on Blood Pressure and Vascular funtion-a Six-month Randomized, Double-blind and Placebo-controlled Trial Among Equol Non-producers of Postmenopausal Women With Prehypertension or Untreated Stage 1 Hypertension
Brief Title: Equol Supplementation on Blood Pressure and Vascular Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Liu Zhaomin, Research Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 471213; CRE-2013.119-T (Other: Ethics Committee of the Chinese University of Hong Kong)
Record Dates: First submitted 2015-07-31; First posted 2015-08-05 (Estimated); Last update posted 2015-08-05 (Estimated); Status verified 2015-08

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- High equol (Active Comparator): High equol group will be given natural S-equol supplementation 20mg per day for 24 week.
  Interventions: Dietary Supplement: High equol group
- Low equol (Active Comparator): Low equol group will be given natural S-equol supplementation 10mg/d (+10mg starch) for 24 weeks
  Interventions: Dietary Supplement: Low equol group
- Placebo (Placebo Comparator): Placebo group will be given placebo control (made from starch) 20 mg per day for 24 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: High equol group — Participants will be give natural S-equol 20mg/d for 24 weeks.
  Arms: High equol
Dietary Supplement: Low equol group — Participants will be give natural S-equol 10mg/d for 24 weeks.
  Arms: Low equol
Dietary Supplement: Placebo — Participants will be give placebo for 24 weeks.
  Arms: Placebo

SUMMARY:
We propose to perform a 24-week randomized, double-blind a placebo-controlled trial among 207 non-equol producing postmenopausal women with prehypertension to examine the effectiveness of equol (10mg and 20mg/d) on 24h ambulatory blood pressure, vascular function and other cardiovascular risks (lipid profile, glycemic control and inflammatory biomarkers) and explore the optimal dosage of equol.

DETAILED DESCRIPTION:
Inclusion criteria

1. Hong Kong Chinese women aged 45-65 y with 2~8 years menopausal;
2. Mean SBP above 130 mmHg or DBP above 80 mmHg or both based on an average of 6 BP readings on two different occasions measured by sphygmomanometer.
3. Equol non-producer is defined as 24-hour urinary log10 S-equol:daidzein ratio less than -1.75 after daidzein challenge (60mg daidzein daily for 7 consecutive days).

Exclusion criteria

1. Subjects on anti-hypertensive medication or with average SBP≥160 or DBP≥100 or both;
2. Use of medications known to affect BP within past 6 months;
3. Medical history or presence of certain chronic diseases that could affect BP or limit the individual's ability to participate in the study;
4. Present or history of certain cancers;
5. Regular smoker or alcohol consumption more than 30 g/day;
6. Known soy allergy.

ELIGIBILITY:
Inclusion Criteria:

1. Hong Kong Chinese women aged 45-65 y with 2~8 years menopausal;
2. mean SBP above 130 mmHg or DBP above 80 mmHg or both based on an average of 6 BP readings on two different occasions measured by sphygmomanometer.
3. Equol non-producer is defined as 24-hour urinary log10 S-equol:daidzein ratio less than -1.75 after daidzein challenge (60mg daidzein daily for 7 consecutive days).
4. Written informed consent will be obtained from all the participants prior to enrolment.

Exclusion Criteria:

1. Subjects on anti-hypertensive medication or with average SBP≥160 or DBP≥100 or both;
2. use of medications known to affect BP within past 6 months (hormone therapy, hypoglycemic or weight reduction agents);
3. medical history or presence of certain chronic diseases (stroke, cardiac infarction, severe liver and renal disease etc.) that could affect BP or limit the individual's ability to participate in the study;
4. present or history of breast cancer, endometrial cancer, ovarian cancer, thyroid disorder, abnormal uterine bleeding after menopause;
5. regular smoker or alcohol consumption more than 30 g/day;
6. known soy allergy.

Ages: 48 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 207 (Estimated)
Dates: Start 2015-10; Primary Completion 2018-07 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Ambulatory blood pressure | 24 weeks

REFERENCES:
- [Derived] Liu ZM, Ho SC, Chen YM, Xie YJ, Huang ZG, Ling WH. Research protocol: effect of natural S-equol on blood pressure and vascular function--a six-month randomized controlled trial among equol non-producers of postmenopausal women with prehypertension or untreated stage 1 hypertension. BMC Complement Altern Med. 2016 Mar 1;16:89. doi: 10.1186/s12906-016-1065-5. PMID 26928904